CLINICAL TRIAL: NCT06595485
Title: Development of Online Mindfulness-Based Intervention for Thai-Depressed Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mae Fah Luang University (Other)
Responsible Party: Principal Investigator, Chuntana Reangsing, Principle investigator, Mae Fah Luang University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Mae Fah Luang Unviersity_002
Record Dates: First submitted 2024-08-27; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Depression in Adolescence
Keywords: depression; Mindfulness; psychological well being; Quality of life
MeSH Terms: conditions — Depression; Psychological Well-Being

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: we will collected outcomes via online application
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- online mindfulness -base intervention (Experimental)
  Interventions: Behavioral: online mindfulness based intervention
- waitlist control group (No Intervention)

INTERVENTIONS:
Behavioral: online mindfulness based intervention — We anticipate the online MBI to be 10-20 minutes once daily, at least 5 days per week, for 8 weeks. Online MBI will be available free of charge on iOS and Android platforms. Participants will be instructed to download the app and use for practices. The online MBI group will be introduced to practice including mindful breathing (simple attention to the flow of the breath, inhalations, and exhalations), body scan (attention and awareness of different body parts) and practice of non-judgement of thoughts and emotions and guided meditation (sitting meditation). In addition, we anticipate participants in MBI group will have a group discussion via skype, 30 minute a week for 8 weeks. Moreover, we anticipate participants in MBI group to record how they practice in each day (attendance) as home assignment using online MBI application. For the details of mindfulness practice, we will develop based on data from interview and focus group
  Arms: online mindfulness -base intervention

SUMMARY:
Project: "Development of Online Mindfulness-Based Intervention for Thai-Depressed Adolescents"

For this project we adopted Kabat-Zinn's definition of mindfulness as the intentional and non-judgmental awareness of thoughts, feelings, and sensations that specifically occur in the present moment (Kabat-Zinn, 2003). We hope to help depressed Thai adolescents begin to develop mindfulness as part of their habitual attention and hone present-moment awareness through mindfulness practicing. For their practice, they will be taught to maintain an awareness of their thoughts, emotions, and physical sensations, and relate these to the negative thoughts that typically contribute to the onset of their depression. We believe this will help Thai adolescents better understand the relationship between their thoughts and their depressive symptoms. Once they understand these relationships, their practice will help them become more flexible, reasonable, and positive.

This project will consist of two phases. Phase I: Using the established literature and qualitative interviews and focus groups, we will design, and pilot test an online MBI. In Phase II, we will evaluate the effectiveness of the online MBI by randomizing depressed Thai adolescent volunteers into one of two groups: an online MBI (intervention group) and a usual care waitlist control group (N=182). Depression, grade, well-being, and mindfulness will be measure at four-time points; baseline, immediately post-intervention, and 3- and 6-months post-intervention

DETAILED DESCRIPTION:
Phase I: To develop and pilot test an online mindfulness-based intervention.

* 10 depressed adolescents for in-depth interviews and 10 stakeholders (2 teachers, 3 school health providers/nurses, 2 mental health and psychiatric instructors, and 3 parents of adolescents) for focus groups to develop and customize the online MBI to adolescents.
* 20 depressed adolescents, randomized to two groups (10 each), to pilot test the study for phase II.

Phase II: To evaluate the effects of the online MBI on depressive symptoms, mindfulness, grade, and well-being among depressed Thai adolescents.

* Quantitative sample: 182 Thai-adolescents with depression randomized to two groups (91 each), to test the effectiveness and efficacy of the online MBI.
* Qualitative sample: 20 Thai adolescents with depression for in-depth interview and focus group to get the adolescents' perceptions of the effectiveness of the online MBI.

ELIGIBILITY:
Inclusion Criteria:

We will include adolescents who

1. are between 12 to 20 years of age;
2. have depressive symptoms (the Children Depressive Inventory [CDI] Score >15);
3. are proficient in Thai;
4. have smartphone with iOS/android platform, and
5. volunteer

Exclusion Criteria:

We will exclude adolescents if they have:

1. current presence of physical or mental conditions, such as learning disorders, major depressive disorders (MDD), bipolar disorders, and drug addiction or abuse, all of which make full participation in all aspects of this study questionable,
2. regularly practiced of MBI within the past six months, and
3. lack of access to online MBI application or to Skype technology for online discussion group

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 182 (Actual)
Dates: Start 2022-01-19 (Actual); Primary Completion 2023-01-19 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
the Children's Depression Inventory (CDI)-Thai version | up to 8 weeks
  a self-reported questionnaire. The scale comprises 27 items with 3-point answers to represent level of depression over the last 2 weeks ago. Participants will rate themselves based on how they feel and think, which each statement being identified with a scale from 0 to 2. A score of 15 or higher is generally accepted to reflect a person who has depression (cut point). Participants will take approximately 10-20 minutes to complete the CDI. The CDI has been widely used among Thai populations with support for validity and good internal consistency (Alpha Cronbach = 0.82, Reangsing, 2011)
the Psychological Well-Being Scale-Thai-version | up to 8 weeks
  PWB-S, is developed by Ryff (1989) and back-translation by Klainin-Yobas et al. (2020). The scale is comprised of 18 items with 6 subscales including autonomy, environmental mastery, purpose of life, personal growth, positive relations with other, and self-acceptance. Participants will rate themselves based on how they feel and perception, which each item ranging from (1) strongly disagree to (6) strongly agree. Possible scores are range from 18 to 108, with higher scores indicating psychological well-being. This scale has support for validity and acceptant reliability (Alpha Cronbach=.70-.85, Klainin-Yobas et al., 2020)
the Five-Facets Mindfulness Questionnaires (FFMQ) | up to 8 weeks
  using the Five-Facets Mindfulness Questionnaires (FFMQ) which is a self-report instrument developed by Baer et al. (2008). This scale consists of 39 items, with 5 sub-domains of mindfulness including observing, describing, acting with awareness, nonjudging of inner experience, and nonreactivity to inner experience. Participants will rate each statement with a number that best describes themselves as scale from never or very rarely true (1) to very often or always true (5). The total FFMQ can be divided by 39 to get an average score of mindfulness (Baer et al., 2006). Higher score indicates high of mindfulness level. This scale has been used among Thai people with a good reliability (Alpha Cronbach = .93, Rattanaphet et al., 2016)

CONTACTS AND LOCATIONS:
Locations (1):
- Mae Fah Luang University, Muang Chiangrai, Chiangrai, Thailand

IPD SHARING:
Plan to Share IPD: No
Prohibited from law